CLINICAL TRIAL: NCT06652542
Title: Asthma Exacerbations & Respiratory Management: an International Online Survey Endorsed by the International Association of Non-invasive Ventilation & International College of Experts
Brief Title: Asthma Exacerbations & Respiratory Management International Survey
Acronym: AERMIS
Status: Enrolling by invitation | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Mohammed Hashem Hamza Ahmed, M.D. , Lecturer of Pulmonology, Department of Chest Diseases and Tuberculosis, Assiut University, Assiut University
Other Study IDs: International Asthma Survey
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute Asthma Exacerbations
Keywords: Asthma Exacerbations; International Survey; Attitudes and Preferences; International Association of Non-invasive Ventilation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Asthma is a chronic health condition that affects 300 million humans worldwide and is thought to cause around 1.000 deaths per day. It's estimated that asthma leads to a significant increase in disability adjusted life years (DALYs). Acute asthma exacerbations affect 25-56% of patients with asthma and represent 8% of intensive care unit (ICU) admissions. Acute asthma exacerbations continue to burden different health systems, particularly emergency units and intensive care units, despite vast advances in pharmacological treatment of asthma, development of evidence-based clinical practice guidelines to improve care of asthma.

This alarming situation indicates non-consensus regarding the best approach for managing acute exacerbations of asthma. Despite that variations in clinical practice regarding diagnosis, prevention, education, long-term management and symptom control of asthma have been thoroughly studied globally, less light has been shed on divergence of physicians' approaches when encountering asthmatic patients during acute exacerbations.

DETAILED DESCRIPTION:
Aim of the Study:

Exploring the physicians' knowledge, attitude and current clinical, pharmacological and ventilatory management practices for acute asthma exacerbations.

Methodology:

Study Design:

The survey is intended to be a cross-sectional survey study.

Time Period:

February 2024-February 2025.

Study Settings:

Respondents are to be recruited by the authors, who are to distribute the online survey to targeted colleagues within the medical institutions the authors are affiliated to, and through different national and international scientific societies of common interest in pulmonology and critical care medicine. Individual physicians are free to distribute the online questionnaire form via electronic communication through the channels they deem most appropriate.

Target Respondents:

Physicians involved in the care of adult asthmatic patients (general practitioners, family medicine doctors, internists, pulmonologists, intensivists in different medical ICUs).

Development of the Questionnaire Questions:

First, a thorough revision of existing literature related to different aspects of management of asthma exacerbations was performed. A total of 45 articles published in national and international journals -including review articles, clinical trials, editorials, and meta-analyses-discussing diagnosis, severity assessment, pharmacological and ventilatory management, as well as outcomes of acute asthma exacerbations were examined to find points of variation in clinical practice, distinguish which approaches are evidence-based, and the magnitude and the pattern of deviation from clinical practice guidelines in different countries. Then, data to be explored were organized into seven domains:

Domain 1.: Respondents' characteristics:

This includes age, geographic region, specialty, years of experience, clinical position and academic degree (if present), affiliation, as well as the level of the health care facility through which a respondent provides care to patients presenting with acute asthma exacerbations.

Domain 2.: Diagnosis of acute asthma exacerbations:

Respondents are to report whether their reliance is wholly on clinical judgement or on tools provided by certain local or international practice guidelines when it comes to identifying asthma patients in acute exacerbations and deciding upon emergency room (ER) admission or ICU referral.

Domain 3.: Pharmacological Management of Acute Asthma Exacerbations:

This domain aims to measure the respondents' knowledge about different pharmacological therapies administrated during acute asthma exacerbations, their usual practice as governed by local policies and resources, as well as their individual preferences towards certain approaches, to detect gaps between knowledge and practice. Drugs including bronchodilators, systemic steroids, antibiotics, and anti-histaminic are to be inquired about regarding frequency of use, method of administration, prescribed doses, and ideal/preferred alternatives. Use of other drugs like magnesium sulphate, theophylline, epinephrine, inhaled anesthetics and intravenous ketamine is to be verified, and respondents are asked to report their knowledge about whether the use of any of these drugs is endorsed by any clinical practice guidelines they are aware of.

Domain 4.: Oxygen therapy during acute asthma exacerbations:

This domain screens the knowledge of the respondents about indications of oxygen administration during acute asthma exacerbations, explores their attitude towards the choice of oxygen delivery system. Familiarity of respondents with the settings of high-flow nasal cannula (HFNC), barriers towards its use, as well as physicians' preferences regarding HFNC are also explored.

Domain 5.: Non-invasive ventilation (NIV) in acute asthma exacerbations:

Access to NIV, frequency of its use, the available NIV devices, and the preferred NIV mode and interfaces by a respondent are inquired about. Respondents' knowledge of the physiological rationales behind using NIV, the appropriate settings of NIV for patients presenting with acute asthma exacerbations, and how to address the main problems arising in such patients are challenged. Knowledge, attitudes and respondents' preferences towards use of sedation during NIV in critically ill asthmatics, knowledge of the best approach to deliver nebulized drugs during NIV, understanding of NIV interference with nebulization therapy, as well as individual preferences regarding the method of delivery are all explored. Barriers to the use of NIV for acute asthma exacerbations, and potential complications associated with its application are also investigated.

Domain 6.: Invasive mechanical ventilation (IMV)in acute asthma exacerbations:

Respondents are inquired about frequency of application of IMV in acute asthma exacerbations, the units where IMV is provided, their knowledge about pathophysiology of severe asthma exacerbations, the appropriate mode and settings of MV, the role of sedation and neuromuscular blockade and the respondents' attitudes and preferences towards the use of these drugs and monitoring patients whilst administration of these drugs are explored. Adjustment of ventilatory settings prior to administration of nebulized drugs and frequency of complications during IMV of acute asthma exacerbations are inquired about as well.

Domain 7.: Outcomes of acute asthma exacerbations:

Respondents' knowledge about possible predictors of prognosis of patients presenting with asthma exacerbations is assessed.

Ethical Considerations:

No ethical approval by certain medical ethics commissions is required for this study. However, the online questionnaire form includes a consent statement at the start of the questionnaire that states a declaration of consent and that the respondent is a medical doctor who holds at least a graduate degree in medical science. Answering "yes" leads the respondent to the first domain, while answering "no" automatically leads the respondent to the end of the form to be submitted.

Data Storage and Confidentiality:

Contact information, i.e. e-mail address is set to be optional. Other personal information such as age, years of experience and affiliation are to be collected for the descriptive purposes and depiction of general characteristics of the respondents providing information but are not to be unlawfully shared or distributed. Access to such information is set to be exclusively restricted to the authors of the questionnaire form. After data analysis, results will be published -maintaining respondents' anonymity- and will be available upon request.

Management of Adverse Events:

Given the commitment of the authors to respondents' confidentiality, no adverse events are expected from this study.

Statistical Analysis:

A certified epidemiologist statistician is to help with statistical analysis. Descriptive statistics will be conducted as well as relevant inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

* All practicing physician who may encounter patients with asthma during their clinical practice are invited to participate.

Exclusion Criteria:

* Non-practicing undergraduate medical students

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonologists, internists, paediatricians, and intensivists at primary, secondary, or tertiary health care facility, from different countries and geographic territories, with varying years of experience and academic backgrounds
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Physicians Knowledge & Attitudes: Diagnosis of Asthma Exacerbations | Through study completion i.e. over an average of 1 year
  A respondent chooses from multiple choices a statement that best describes their knowledge/attitudes regarding the criteria used for diagnosis of acute asthma exacerbations (prespecified criteria derived from clinical practice guidelines or local policies rather than clinical judgement) . The number of responding physician to each statement is to be recorded.
Physicians' Knowledge and Attitudes: Pharmacological Management | Through study completion i.e. over an average of 1 year
  A respondent chooses from multiple choices a statement that best describes their knowledge/attitudes regarding the use of different asthma medications (bronchodilators, steroids, sedatives, neuromuscular blockers). The number of responding physician to each statement is to be recorded.
Physicians Knowledge & Attitudes: Ventilatory Management | Through study completion i.e. over an average of 1 year
  A respondent chooses from multiple choices a statement that best describes their knowledge/attitudes regarding the frequency of use of different ventilatory support methods (oxygen therapy, high-velocity nasal insufflation (HVNI), noninvasive ventilation (NIV), invasive mechanical ventilation (IMV)) and the appropriate settings. Physicians' awareness about expected adverse events of each modality is tested. The number of responding physician to each statement is to be recorded.

SECONDARY OUTCOMES:
Physicians' Knowledge: Prognosis of Acute Asthma Exacerbations | Through study completion i.e. over an average of 1 year
  A respondent chooses from multiple choices the predictors they think are predictors of poor asthma outcomes, according to their current state of knowledge. The number of responding physician to each statement is to be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M. Esquinas, PhD, FCCP, Study Director — International Council Respiratory Care, ICU, Hospital Morales Meseguer, Murcia, Spain.; Mohammed M. Metwally, PhD, FCCR, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention,2024. Updated May 2024.
- [Background] Wang Z, Li Y, Gao Y, Fu Y, Lin J, Lei X, Zheng J, Jiang M. Global, regional, and national burden of asthma and its attributable risk factors from 1990 to 2019: a systematic analysis for the Global Burden of Disease Study 2019. Respir Res. 2023 Jun 23;24(1):169. doi: 10.1186/s12931-023-02475-6. PMID 37353829
- [Background] Wang E, Wechsler ME, Tran TN, Heaney LG, Jones RC, Menzies-Gow AN, Busby J, Jackson DJ, Pfeffer PE, Rhee CK, Cho YS, Canonica GW, Heffler E, Gibson PG, Hew M, Peters M, Harvey ES, Alacqua M, Zangrilli J, Bulathsinhala L, Carter VA, Chaudhry I, Eleangovan N, Hosseini N, Murray RB, Price DB. Characterization of Severe Asthma Worldwide: Data From the International Severe Asthma Registry. Chest. 2020 Apr;157(4):790-804. doi: 10.1016/j.chest.2019.10.053. Epub 2019 Nov 27. PMID 31785254
- [Background] Mohamed AZELA, Shaaban LH, Gad SF, Azeem EA, Gamal Elddin W. Acute severe asthma in emergency department: clinical characteristics, risk factors, and predictors for poor outcome. The Egyptian Journal of Bronchology. 2022;16(1).
- [Background] Gayen S, Dachert S, Lashari BH, Gordon M, Desai P, Criner GJ, Cardet JC, Shenoy K. Critical Care Management of Severe Asthma Exacerbations. J Clin Med. 2024 Feb 1;13(3):859. doi: 10.3390/jcm13030859. PMID 38337552
- [Background] Aggarwal B, Al-Moamary M, Allehebi R, Alzaabi A, Al-Ahmad M, Amin M, Damayanti T, Van Tho N, Quyen PTL, Sriprasart T, Poachanukoon O, Yu-Lin AB, Ismail AI, Limpin MEB, Koenig S, Levy G, Phansalkar A, Rafih F, Silvey M, Miriams L, Milligan G. APPaRENT 3: Asthma Patients' and Physicians' Perspectives on the Burden and Management of Asthma in Seven Countries. Adv Ther. 2024 Aug;41(8):3089-3118. doi: 10.1007/s12325-024-02900-2. Epub 2024 Jun 14. PMID 38874879
- [Background] Garcia-Marcos L, Chiang CY, Asher MI, Marks GB, El Sony A, Masekela R, Bissell K, Ellwood E, Ellwood P, Pearce N, Strachan DP, Mortimer K, Morales E; Global Asthma Network Phase I Study Group. Asthma management and control in children, adolescents, and adults in 25 countries: a Global Asthma Network Phase I cross-sectional study. Lancet Glob Health. 2023 Feb;11(2):e218-e228. doi: 10.1016/S2214-109X(22)00506-X. PMID 36669806
- [Background] Ibrahim AO, Aremu SK, Afolabi BA, Ajani GO, Kolawole FT, Oguntoye O. Acute severe asthma and its predictors of mortality in rural Southwestern Nigeria: a-five year retrospective observational study. Chron Respir Dis. 2023 Jan-Dec;20:14799731221151183. doi: 10.1177/14799731221151183. PMID 36652901
- [Background] Selroos O, Kupczyk M, Kuna P, Lacwik P, Bousquet J, Brennan D, Palkonen S, Contreras J, FitzGerald M, Hedlin G, Johnston SL, Louis R, Metcalf L, Walker S, Moreno-Galdo A, Papadopoulos NG, Rosado-Pinto J, Powell P, Haahtela T. National and regional asthma programmes in Europe. Eur Respir Rev. 2015 Sep;24(137):474-83. doi: 10.1183/16000617.00008114. PMID 26324809
- [Background] Mortimer K, Reddel HK, Pitrez PM, Bateman ED. Asthma management in low and middle income countries: case for change. Eur Respir J. 2022 Sep 15;60(3):2103179. doi: 10.1183/13993003.03179-2021. Print 2022 Sep. PMID 35210321
- [Background] Talbot T, Roe T, Dushianthan A. Management of Acute Life-Threatening Asthma Exacerbations in the Intensive Care Unit. Applied Sciences. 2024;14(2)
- [Background] Zeitouni MO, Al-Moamary MS, Coussa ML, Riachy M, Mahboub B, AlHuraish F, Zidan MH, Metwally MM, Aksu K, Yavuz E, Kalla IS, Chakaya J, Abdelmadjid S, Ghedira H. Challenges and recommendations for the management of asthma in the Middle East and Africa. Ann Thorac Med. 2022 Apr-Jun;17(2):71-80. doi: 10.4103/atm.atm_469_21. Epub 2022 Apr 19. PMID 35651897
- See also: The online questionnaire form distributed for recruiting respondents — https://docs.google.com/forms/d/e/1FAIpQLSeRO5cwZRfYSd5EmWYTq4GEFblx04YK-WdeGJXCKgHO9v28HA/viewform?usp=pp_url